CLINICAL TRIAL: NCT01714102
Title: The Effects of Trans-Resveratrol (RSV) on Insulin Resistance, Inflammation, and the Metabolic Syndrome: A Placebo Controlled, Double-Blind Study.
Brief Title: Resveratrol and the Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Principal Investigator, Jeanne Walker, Senior Clinical Nurse Practitioner & Research Coordinator, Rockefeller University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JWA-0786
Record Dates: First submitted 2012-10-16; First posted 2012-10-25 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Obesity; Insulin Resistance; Metabolic Syndrome
Keywords: Obesity; Insulin resistance; Metabolic syndrome; Pre-diabetes
MeSH Terms: conditions — Obesity; Insulin Resistance; Metabolic Syndrome; Glucose Intolerance | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo for 30 days
  Interventions: Dietary Supplement: Resveratrol
- Resveratrol (Active Comparator): 1000 mg PO BID for 30 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo manufactured to mimic resveratrol tablet
  Arms: Resveratrol
Dietary Supplement: Resveratrol — Resveratrol PO BID for 30 days
  Arms: Placebo

SUMMARY:
Metabolic syndrome is a serious health condition that affects about 35 percent of adults and places them at higher risk of cardiovascular disease, diabetes, stroke and diseases related to fatty buildups in artery walls. The underlying causes of metabolic syndrome are obesity, being overweight, physical inactivity and genetic factors. In recent decades, the prevalence has increased dramatically in the United States. Lifestyle interventions including dietary modification, physical activity and weight loss form the basis of treatment for these patients. However, research has shown that even when people are able to incorporate these changes, they often revert back to their usual lifestyle resulting in weight gain and continued risk for diabetes and heart disease.

Resveratrol, a natural plant derived compound found in grapes, peanuts and red wine, has been found to reverse some of the features of the metabolic syndrome (insulin resistance, high triglycerides, high blood pressure) in rodents. These improvements occurred without weight loss, and were proven to be a direct result of resveratrol ingestion. Other studies reveal improvement in cardiovascular health, tumor suppression, and longevity. However, there are few studies investigating these beneficial effects in humans. Investigators propose to prove that resveratrol, administered to subjects with the metabolic syndrome, under controlled conditions of weight stability, common diet, and strict compliance with the study drug, will improve the symptoms of the metabolic syndrome, thereby decreasing the chance of developing diabetes or heart disease.

DETAILED DESCRIPTION:
The metabolic syndrome is a serious health condition that affects about 35 percent of adults and places them at higher risk of cardiovascular disease, diabetes, stroke and diseases related to fatty buildups in artery walls. The underlying causes of metabolic syndrome are obesity, being overweight, physical inactivity and genetic factors. In recent decades, the prevalence has increased dramatically in the United States. Lifestyle interventions including dietary modification, physical activity and weight loss form the basis of treatment for these patients. However, research has shown that even when people are able to incorporate these changes, they often revert back to their usual lifestyle resulting in weight gain and continued risk for diabetes and heart disease.

Resveratrol, a natural plant derived compound found in grapes, peanuts and red wine, has been found to reverse some of the features of the metabolic syndrome (insulin resistance, high triglycerides, high blood pressure) in rodents. These improvements occurred without weight loss, and were proven to be a direct result of resveratrol ingestion. Other studies reveal improvement in cardiovascular health, tumor suppression, and longevity. However, there are few studies investigating these beneficial effects in humans. In a systematic review of resveratrol research, the authors conclude that "in contrast to the lacking data of resveratrol in humans, the animal data are promising and indicate the need for further human clinical trials." Of the small clinical studies that have been done, the results are encouraging. Improvement in triglycerides, blood pressure and insulin resistance were noted. Resveratrol was well tolerated without serious side effects. These studies, however, did not recruit subjects with the metabolic syndrome, nor were they tightly controlled.

The investigators propose to prove that resveratrol, administered to subjects with the metabolic syndrome, under controlled conditions of weight stability, common diet, and strict compliance with the study drug, will improve the symptoms of the metabolic syndrome, thereby decreasing the chance of developing diabetes or heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 - 60 year old men
* Willingness to be randomized to resveratrol or placebo.
* BMI 30-40
* Evidence of insulin resistance with one of the following:

  2 hr oral glucose tolerance result =/>120mg/dl at 2hrs acanthosis nigricans, or HgA1C 5.7 - 7.9%, or FBS >/= 100 mg/dl AND at least 2 of the following: waist circumference > 102 cm triglycerides > 150 but < 500 mg/dL HDL < 40 mg/dL Pre- hypertension or hypertension: BP>120/80 mmHg but <150/90 mmHg
* Willingness to consume only study food and drink during the in-pt phases
* Willingness to avoid the use of over-the-counter medications, herbs, or supplements within the last 30 days.
* Willingness to avoid NSAIDS (advil, aleve, motrin, etc.) and aspirin for the entire study
* Willingness to avoid ingestion of any foods containing peanuts, bilberries, blueberries, cranberries, strawberries, raspberries, grapes, grape juice, cocoa powder, dark chocolate, and red wine throughout the entire study, including run-in period.
* Willingness to maintain weight for the duration of the study.
* Willingness not to start an exercise regime during study participation

Exclusion Criteria:

* Tobacco smoker any time within the last 3 months
* Bleeding disorder by history or by Bleeding Questionnaire results
* History, physical or EKG findings suggestive of CV disease including angina, MI, hx of med/surg tx of atherosclerotic heart disease, or congestive heart disease
* BP > 145/90 after 10 minutes of rest on 2 or more screening visits
* Fasting glucose > 165 mg/dL at screening
* HbA1C > 8.0 at screening
* Current use of oral hypoglycemic agents
* Chronic glucocorticosteroid use or use of oral glucocorticosteroids for 5 days within the last year (inhaled glucocorticosteroid use may be acceptable; this will be determined by the PI)
* Current use of over the counter or prescription weight loss medication
* Current use or within the last 30 days, any cholesterol lowering medications (statins, fibrates, red yeast rice, niacin).
* Hyperthyroidism or untreated hypothyroidism
* Obstructive sleep apnea, or significant symptoms suggestive of this condition.
* Current use of anticoagulants
* Known history of chronic hepatitis or liver enzymes (ALT or AST > 2.5 times the normal upper limit)
* Known HIV infection or confirmed positive test for HIV antibodies at screening
* Inflammatory bowel disease
* Active cancer (currently under treatment)
* Other medical condition that may cause significant weight loss or gain
* Chronic or acute renal disease
* Seizure disorder
* History of any psychiatric hospital admission within the last 2 years
* History of schizophrenia, psychosis, or bipolar disease
* History, physical, social or lab findings suggestive of any medical or psychological condition that would, in the opinion of the PI, impact the subject's ability to successfully participate in the study.
* Alcohol or drug abuse within the last 2 years
* Any medications metabolized by cytochrome p450 3A4 (CYPA3A4) (see attachment of these medications as an appendix)
* Any autoimmune disease (ie rheumatoid arthritis, systemic lupus erythematosis, psoriasis)
* Physical condition requiring special diet (ie celiac disease)

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Reduction in Insulin resistance | Days 4-8 and Days 31-35
  Investigators anticipate resveratrol will have positive effect (ie reduction) on Insulin resistance as determined by Euglycemic hyperinsulinemic clamp

SECONDARY OUTCOMES:
Reduction in serum cytokines/chemokines | Days 4-8 and Days 31-35
  Investigators anticipate resveratrol will have positive effect (ie reduction) on Serum cytokines/chemokines: IL6, IL10, TNFalpha, hsCRP, leukocytes, PAI-1, fibrinogen, adiponectin, MCP-1,GLP-1, leptin, insulin, serum endotoxins
Reduction in blood pressure measurements | Days 4-8 and Days 31-35
  24 hour systolic blood pressure measurements
Reduction lipid values | Days 4-8 and Days 31-35
  Lipid values to be reviewed: cholesterol, LDL, HDL, TG
Reduction in crown like structures and adipose tissue mass | Days 4-8 and Days 31-35
  Crown like structures in adipose tissue, and adipose tissue mass
Changes in HOMA-IR | Days 4-8 and Days 31-35
  Changes in 2 hr oral glucose tolerance test HOMA-IR
Changes in gene expression in adipose tissue | Days 4-8 and Days 31-35
  Changes in RNA sequencing of adipose tissue
Changes in gene expression in stool | Days 4-8 and Days 31-35
  Changes in microbiome and RNA gene expression in stool samples

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Walker, MSN/NP-C, Principal Investigator — The Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States